CLINICAL TRIAL: NCT03814798
Title: A Multicenter, Randomized, Cross-over, Open-label Study to Evaluate IGSC 20% Flexible Dosing Including Daily Push Dosing In Treatment-Experienced Subjects With Primary Immunodeficiency (PI) and Evaluation of Loading/Maintenance IGSC 20% in Treatment-Naïve Subjects With PI
Brief Title: Study Evaluating IGSC 20% Flexible Dosing in Treatment-Experienced and Treatment-Naive Subjects With Primary Immunodeficiency
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the regulatory approval of the product in this indication, a large portion of the study becomes unnecessary.
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GC1701
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): IGSC 20% daily push versus every 2 weeks pump or the reverse sequence
  Interventions: Biological: IGSC 20% daily push versus every 2 weeks pump
- Cohort 2 (Experimental): IGSC 20% daily push versus once a week pump or the reverse sequence
  Interventions: Biological: IGSC 20% daily push versus once a week pump
- Cohort 3 (Experimental): IGSC 20% daily push versus 2 times per week pump or the reverse sequence
  Interventions: Biological: IGSC 20% daily push versus 2 times per week pump
- Treatment-Naive IGSC 20% pump dosing (Experimental): IGSC 20% 150 mg/kg
  Interventions: Biological: IGSC 20% 150 mg/kg

INTERVENTIONS:
Biological: IGSC 20% daily push versus every 2 weeks pump — IGSC 20% syringe daily push dosing for 16 weeks followed by every 2 weeks pump dosing for 16 weeks or the reverse sequence
  Arms: Cohort 1
Biological: IGSC 20% daily push versus once a week pump — IGSC 20% syringe daily push dosing for 16 weeks followed by once weekly ambulatory pump administration dosing for 16 weeks or the reverse sequence
  Arms: Cohort 2
Biological: IGSC 20% daily push versus 2 times per week pump — IGSC 20% syringe daily push dosing for 16 weeks followed by 2 times/week ambulatory pump administration on preselected days (eg, Monday and Thursday) not less than 3 days apart for 16 weeks or the reverse sequence
  Arms: Cohort 3
Biological: IGSC 20% 150 mg/kg — loading dose of IGSC 20% consisting of 5 consecutive daily doses of 150 mg/kg/day (Week 0, Days 1-5) followed by weekly infusions of IGSC 20% 150 mg/kg starting Week 1 (Day 8) through Week 32 using an infusion SC pump
  Arms: Treatment-Naive IGSC 20% pump dosing

SUMMARY:
This is a prospective, multi-center, randomized, open-label, 2-period cross-over study (16 weeks per treatment period) to evaluate flexible dosing and daily push dosing of IGSC 20% in treatment-experienced subjects with PI. An additional, separate cohort of treatment-naïve, non-randomized subjects who will not be part of the crossover are included and will receive a loading dose of 5 consecutive daily doses of IGSC 20% followed by weekly infusions of IGSC 20% starting Week 1 (Day 8) through Week 32 (end of Treatment Phase).

For treatment-experienced subjects, the study consists of a Screening Visit, Baseline Visit, 16-week Treatment Period 1, 16-week Treatment Period 2, and Final Visit/Early Termination Visit. For treatment-naïve subjects, the study consists of a Screening Visit, a Baseline Visit, a 32-week Treatment Phase, and Final Visit/Early Termination Visit.

Approximately 54 treatment-experienced subjects and approximately 6 treatment-naïve subjects will be enrolled at study centers in the United States (US) and European Union (EU).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, open-label, 2-period cross-over study (16 weeks per treatment period) to evaluate flexible dosing and daily push dosing of IGSC 20% in treatment-experienced subjects with PI. There is an additional, separate cohort of treatment-naïve, non-randomized subjects with PI who will not be part of the crossover.

Treatment-experienced subjects entering the study will maintain the same IgG dose (mg/kg) received prestudy that will be normalized to the study-assigned dose-time interval (ie, there will be 1:1 correspondence regardless of prestudy route of administration [intravenous [IV] or SC]). Treatment-experienced subjects will be randomized in a 1:1:1 ratio into 1 of 3 parallel cohorts consisting of 18 subjects each as follows:

Cohort 1 (daily push compared with every 2 weeks [biweekly] pump) will evaluate syringe daily push dosing versus every 2 weeks [biweekly] ambulatory pump administration. Subjects will be randomized in a 1:1 ratio to 1 of 2 sequences, either beginning with syringe daily push dosing for 16 weeks and then crossing over to ambulatory pump administration every 2 weeks for 16 weeks or the reverse sequence.

Cohort 2 (daily push compared with once weekly pump) will evaluate syringe daily push dosing versus once weekly ambulatory pump administration. Subjects will be randomized in a 1:1 ratio to 1 of 2 sequences, either beginning with syringe daily push dosing for 16 weeks and then crossing over to ambulatory pump administration once every week for 16 weeks or the reverse sequence.

Cohort 3 (daily push compared with 2 times/week pump) will evaluate syringe daily push dosing versus 2 times/week ambulatory pump administration. Ambulatory pump dosing will take place on preselected days (eg, Monday and Thursday) not less than 3 days apart. The dosing days should remain constant for the duration of the study. Subjects will be randomized in a 1:1 ratio to 1 of 2 sequences, either beginning with syringe daily push dosing for 16 weeks and then crossing over to ambulatory pump administration 2 times/week for 16 weeks or the reverse sequence.

The treatment-naïve cohort will receive a loading dose of 5 consecutive daily doses of IGSC 20% 150 mg/kg/day (Week 0, Days 1-5) followed by weekly infusions of 150 mg/kg starting Week 1 (Day 8) through Week 32 (end of Treatment Phase).

ELIGIBILITY:
Inclusion Criteria:

For treatment-experienced subjects:

* Has documented and confirmed pre-existing diagnosis of PI with features of hypogammaglobulinemia requiring IgG replacement therapy including but not limited to the following humoral-based immunodeficiency syndromes (eg, X-linked agammaglobulinemia, common variable immunodeficiency), and combined immunodeficiency syndromes without lymphocytopenia (eg, hyper immunoglobulin M immunodeficiency syndrome).
* Has not had a SBI or been hospitalized for infection of any etiology (eg, viral, fungal, parasitic) within the last 3 months prior to screening or during screening.
* Is currently receiving IgG replacement therapy for ≥3 months via IV or SC infusion. Subjects receiving IVIG prior to study must receive a dosage of at least 200 mg/kg per infusion
* Has Screening IgG trough levels ≥500 mg/dL. Note: If screening trough levels are not above this threshold, the subjects will be considered a screen failure, but may be rescreened following dose adjustment of their original IgG replacement therapy regimen and maintaining stable dosing for a period of at least 3 months prior to screening a second time.
* Has signed an informed consent. Note: The subject must sign the informed consent form (ICF) if at least 18 years old; for children of younger age, the subject's parent or legal guardian must sign the ICF and if appropriate/applicable, the subject must sign a Child Assent form approved by the IRB/EC per the institution's requirements

For treatment-naïve subjects:

* Has documented and confirmed diagnosis of PI with features of hypogammaglobulinemia requiring IgG replacement therapy including but not limited to the following humoral-based immunodeficiency syndromes (eg, X-linked agammaglobulinemia, common variable immunodeficiency), and combined immunodeficiency syndromes without lymphocytopenia (eg, hyper immunoglobulin M immunodeficiency syndrome).
* Has never received IgG replacement treatment (ie, no prior immune globulin replacement therapy)
* Has Screening IgG level ≤400 mg/dL
* Does not have an SBI nor requires hospitalization for infection of any etiology (eg, viral, fungal, parasitic) during screening or at baseline.
* Has signed an informed consent. Note: The subject must sign the informed consent form (ICF) if at least 18 years old; for children of younger age, the subject's parent or legal guardian must sign the ICF and if appropriate/applicable, the subject must sign a Child Assent form approved by the IRB/EC per the institution's requirements

Exclusion Criteria:

For all subjects:

* Has clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the trial or place the subject at undue medical risk.
* Has had a known serious adverse reaction to immunoglobulin or any anaphylactic reaction to blood or any blood-derived product
* Has a history of blistering skin disease, clinically significant thrombocytopenia, bleeding disorder, diffuse rash, recurrent skin infections, or other disorders where SC therapy would be contraindicated during the study.
* Has known isolated IgG subclass deficiency; isolated specific antibody deficiency (SAD) or selective IgG deficiency; or transient hypogammaglobulinemia of infancy. Note: Subjects are not to be enrolled if their primary PI diagnosis does not entail an actual quantitative deficit in total IgG. For example, SAD is defined as an impaired specific IgG response to pneumococcal vaccine with normal serum concentrations of IgG, IgM, and IgA. Isolated IgG subclass deficiency is defined as an abnormally low level of 1 or more IgG subclass in subjects with normal levels of total IgG and IgM.
* Has known selective IgA deficiency (with or without antibodies to IgA) (Note: exclusion is for the specific diagnostic entity. It does not exclude other forms of humoral primary immunodeficiency which have decreased IgA in addition to decreased IgG requiring IgG replacement).
* Is female of childbearing potential who is pregnant, has a positive pregnancy test at screening (serum human chorionic gonadotropin [HCG]- based assay), is breastfeeding, or is unwilling to practice a highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study. Note: True abstinence: When this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods], declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception.)
* Has significant proteinuria (≥3+ or known urinary protein loss >1 g/24 hours or nephrotic syndrome), has acute renal failure, is on dialysis, and/or has severe renal impairment on Screening laboratory testing (blood urea nitrogen or creatinine more than 2.5 times the upper limit of normal [ULN]).
* Has screening values of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding more than 2.5 times the ULN for the expected normal range for the testing laboratory.
* Has hemoglobin <9 g/dL at screening.
* Has a history (either 1 episode within the year prior to the Screening Visit or 2 previous episodes over a lifetime) of or current diagnosis of thromboembolism (eg, myocardial infarction, cerebrovascular accident or transient ischemic attack) or deep venous thrombosis.
* Is currently receiving anti-coagulation therapy which would make SC administration inadvisable (vitamin K antagonists, nonvitamin K antagonist oral anticoagulants [eg, dabigatran etexilate targeting Factor IIa, rivaroxaban, edoxaban, and apixaban targeting Factor Xa], and parenteral anticoagulants [eg, fondaparinux]).
* Currently has a known hyperviscosity syndrome.
* Has an acquired medical condition that is known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1000/μL [1.0 x 10^9/L]), or human immunodeficiency virus infection/acquired immune deficiency syndrome.
* Has a known previous infection with or clinical signs and symptoms consistent with current hepatitis B virus or hepatitis C virus infection.
* If <18 years of age, has non-controlled arterial hypertension at a level of greater than or equal to the 90th percentile blood pressure (either systolic or diastolic) for their age and height or the adult subject has non- controlled arterial hypertension (systolic blood pressure [SBP] >160 mmHg and/or diastolic blood pressure [DBP] >100 mmHg).
* Is receiving any of the following medications:

  1. immunosuppressants including chemotherapeutic agents;
  2. immunomodulators; (c) long-term systemic corticosteroids defined as daily dose >1 mg of prednisone equivalent/kg/day for >30 days. Note: Intermittent courses of corticosteroids of not more than 10 days would not exclude a subject. Inhaled or topical corticosteroids are allowed.
* Has known substance or prescription drug abuse.
* Has participated in another clinical trial within 30 days prior to screening (observational studies without investigative treatments [non- interventional] are permitted) or has received any investigational blood product with the exception of other IgG products within the previous 3 months.
* Is a subject/caregiver unwilling to comply with any aspect of the protocol, including home SC infusions, blood sampling, and completion of a SC infusion diary for the duration of the study.
* Is a mentally challenged subject who cannot give independent informed consent or assent.
* In the opinion of the investigator, the subject may have compliance problems with the protocol and the procedures of the protocol.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Steady-state mean trough (predose) concentration of total IgG | Baseline to Week 32
  Steady-state mean trough (predose) concentration following SC administration of IGSC 20% in treatment-experienced subjects

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The South Bend Clinic LLP, South Bend, Indiana
  - Optimed Research LTD, Columbus, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No